CLINICAL TRIAL: NCT03117985
Title: Tracking and Exploring the Source of Viral REbound
Acronym: TESOVIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no interesting results
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: Laboratoire de Virologie Moléculaire de Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO 2016-05
Record Dates: First submitted 2017-03-24; First posted 2017-04-18 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Hiv
Keywords: HIV reservoirs; HIV persistence; Viral rebound
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antiretroviral therapy (Experimental): Stopping antiretroviral therapy
  Interventions: Other: no drug

INTERVENTIONS:
Other: no drug — Stopping antiretroviral therapy

SUMMARY:
Phylogenic analysis of viruses hosted in marker positive reservoir cells including CD32a+ CD4 T lymphocytes and rebounding viruses after treatment interruption

ELIGIBILITY:
Inclusion Criteria:

* - Age>18year old
* Nadir CD4>200/mm3
* CD4/CD8 ratio> 0.5
* Continuous antiretroviral therapy for more than 2 years
* Plasma Human Immunodeficiency Virus (HIV) 1 Ribonucleic acid (RNA) <50 copies/ml in the last 2 years
* Viral Load (VL)<20copies at inclusion
* Patients who are willing to participate and who understand the trial (particularly, the obligation to have protected intercourse during the study).
* Informed consent
* Short half-life treatment
* Health insurance
* A subset of CD4 (T4cells) express CD32a.

Exclusion Criteria:

* - Acquired Immune Deficiency Syndom (AIDS)
* Pregnancy
* Human immunodeficiency virus (HIV)-2 co infection
* Thrombopenia
* Neurological events during primary infection
* Hepatitis B + (HBV+)
* Hepatitis C + (HCV+)
* Cancer during the last 5 years.
* Life expectancy < 12 months
* Autoimmunity
* Acute infectious disease in the last 60 days.
* Hemoglobin<7g/dl
* Glomerular filtration < 60ml/min
* Refusing protected intercourse
* Risk of HIV transmission
* Psychiatric disorders.
* Alcool and drug abuse
* Involvement in another clinical trial evaluating a therapeutic.
* Being under tutorship
* Being deprived of liberty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Genetic Cartography | Week 1
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml
Genetic Cartography | Week 2
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml
Genetic Cartography | Week 3
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml
Genetic Cartography | Week 4
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml
Genetic Cartography | Week 5
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml
Genetic Cartography | Week 6
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml
Genetic Cartography | Week 8
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml
Genetic Cartography | Week 10
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml
Genetic Cartography | Week 12
  Measuring the genetic distance between viruses contained in marker positive reservoir cells including CD32a+ CD4 T (T4cells) lymphocytes and viruses rebounding after treatment interruption. This cartography will be made when Plasma Human Immunodeficiency Virus -1 ribonucleic acid (RNA) superior or equal to 1000 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: LAURENT HOCQUELOUX, Study Director — CHR ORLEANS
Locations (1):
- Chr Orleans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Descours B, Petitjean G, Lopez-Zaragoza JL, Bruel T, Raffel R, Psomas C, Reynes J, Lacabaratz C, Levy Y, Schwartz O, Lelievre JD, Benkirane M. CD32a is a marker of a CD4 T-cell HIV reservoir harbouring replication-competent proviruses. Nature. 2017 Mar 23;543(7646):564-567. doi: 10.1038/nature21710. Epub 2017 Mar 15. PMID 28297712